CLINICAL TRIAL: NCT06476808
Title: A Phase 1/1b First-in-human Study of BMS-986463 in Advanced Malignant Tumors
Brief Title: A Study to Evaluate the Safety, Tolerability, and Efficacy of Escalating Doses of BMS-986463 in Participants With Select Advanced Malignant Tumors.
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CA231-0000
Record Dates: First submitted 2024-06-21; First posted 2024-06-26 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-10

CONDITIONS: High-grade Serous Ovarian Carcinoma (HGSOC); Uterine Serous Carcinoma (USC); Non-small Cell Lung Cancer (NSCLC)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1: Dose Escalation (Experimental)
  Interventions: Drug: BMS-986463
- Arm 2: Dose Expansion (Experimental)
  Interventions: Drug: BMS-986463

INTERVENTIONS:
Drug: BMS-986463 — Specified dose on specified days

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, and efficacy of escalating doses of BMS-986463 in participants with select advanced malignant tumors.

ELIGIBILITY:
Inclusion Criteria

* Participants must have an Eastern Cooperative Oncology Group Performance Status of 0 or 1.
* Participants must have at least 1 lesion accessible for biopsy in addition to the target lesion, from which a fresh pre treatment biopsy must be obtained.
* Participants must have an unresectable/metastatic carcinoma.

Exclusion Criteria

* Participants must not have Leptomeningeal metastases.
* Participants must not have concurrent malignancy (present during screening) requiring treatment or history of prior malignancy active within 2 years prior to treatment.
* Participants must not have had any prior radiation therapy within 2 weeks prior to start of study treatment.
* Other protocol-defined Inclusion/Exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2024-09-06 (Actual); Primary Completion 2028-12-19 (Estimated); Study Completion 2028-12-19 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events (AEs) | Up to 108 weeks
Number of participants with serious adverse events (SAEs) | Up to 108 weeks
Number of participants with AEs meeting protocol defined dose-limiting toxicity (DLT) criteria | Up to 108 weeks
Number of participants with AEs leading to discontinuation | Up to 108 weeks
Number of participants with AEs leading to death | Up to 108 weeks

SECONDARY OUTCOMES:
Maximum observed concentration (Cmax) | Up to 104 weeks
Area under the concentration-time curve (AUC) | Up to 104 weeks
Time of maximum observed concentration (Tmax) | Up to 104 weeks
Objective response rate (ORR) | Up to 104 weeks
Disease control rate (DCR) | Up to 104 weeks
Duration of response (DOR) | Up to 104 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (16):
- United States (5):
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - Valkyrie Clinical Trials, Los Angeles, California
  - John Theurer Cancer Center at Hackensack University Medical Center, Hackensack, New Jersey
  - Local Institution - 0045, Columbus, Ohio
  - Local Institution - 0046, Dallas, Texas
- Canada (4):
  - BC Cancer Vancouver, Vancouver, British Columbia
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - Centre Hospitalier de l'Université de Montréal, Montreal, Quebec
  - Jewish General Hospital, Montreal, Quebec
- France (3):
  - Local Institution - 0031, Villejuif, Val-de-Marne
  - Local Institution - 0036, Borddeaux Cedex
  - Local Institution - 0035, Lyon
- Italy (2):
  - Local Institution - 0032, Rozzano, Milano
  - Local Institution - 0033, Milan
- Spain (2):
  - Local Institution - 0041, Avda.Pio XII 36,
  - Local Institution - 0042, Barcelona

IPD SHARING:
Plan to Share IPD: Yes
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria. Additional information regarding Bristol Myer Squibb's data sharing policy and process can be found at: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See plan description
Access Criteria: See plan description
URL: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsclinicaltrials.com/us/en/clinical-trials/NCT06476808.html